CLINICAL TRIAL: NCT03350919
Title: Visual Restoration for Hemianopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Envision Solutions, LLC (Other Government)
Responsible Party: Principal Investigator, Steven Feldon, Professor and Chair of Ophthalmology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69879
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Stroke Induced Vision Loss; Hemianopia; Quadrantanopia
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Training in the blind field (Experimental): Training in the blind field using software
  Interventions: Device: Training in the blind field
- Training in the intact field (Experimental): Training in the intact field using software
  Interventions: Device: Training in the intact field

INTERVENTIONS:
Device: Training in the blind field — A computer software and chin-rest necessary to perform visual training will be loaned to each patient to use at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a pre-determined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. They will train daily (about 40-60 minutes total), 5 to 7 days per week, for at least 24 weeks.
  Arms: Training in the blind field
Device: Training in the intact field — A computer software and chin-rest necessary to perform visual training will be loaned to each patient to use at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a pre-determined location in the intact field of vision. The computer program will automatically create a record of patient performance during each home training session. They will train daily (about 40-60 minutes total), 5 to 7 days per week, for at least 24 weeks.
  Arms: Training in the intact field

SUMMARY:
The purpose of this research is to assess the efficacy of a visual training task on reducing the size of a visual field deficit caused by brain damage in adults, and its ability to improve visual functions in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-75 years old
* Ability and willingness to sign informed consent
* Willingness to participate in both the training and evaluation sessions
* MRI or CT scan demonstrating lesion in the occipital lobe of the brain and/or affecting white matter tracts that provide visual input to the occipital lobe of the brain
* Brain injury due to ischemic or hemorrhagic causes that occurs after age 18 and at least 90 days prior to screening visit
* At least two reliable HVF's demonstrating good fixation and a stable homonymous incomplete (e.g., quadrantanopia or relative defect) or complete hemianopia
* Reliable HVFs with repeat HVFs if randomization takes place more than 4 weeks after screening visit
* A homonymous, contiguous visual deficit measured by the 24-2 HVF to be a minimum of two testing locations high and two testing locations wide, where impaired locations are any that measure a threshold of less than 15 dB.
* Demonstration of good fixation on visual training task - able to fixate the small targets presented as fixation letters reliably for 1000ms with jitter over less than 1 degree of visual angle in any direction away from target edge

Exclusion Criteria:

* Physical, neurological or mental disability that would interfere with study intervention
* Concurrent participation in "vision therapy" other than standard occupational or physical therapy
* Unreliable visual fields on prior testing, indicated by greater than 20% fixation losses, false positives, or false negatives.
* Inability to discontinue medications judged to affect training and/or assessment (e.g., Ritalin, amphetamines, dopamines, or chemotherapeutic agents)
* Physical condition likely to preclude completion of the clinical trial (e.g. end-stage or uncontrolled cancer, uncontrolled epilepsy, or end-stage heart disease)
* Ocular or neurological condition that would interfere with training or assessment (e.g. damage to the optic nerves or lateral geniculate nucleus, any degenerative ocular condition)
* Best corrected vision worse than 20/40
* Impaired foveal Humphrey sensitivity as indicated by the HVF tests.
* Presence of vision loss resulting from ocular disease or disorder
* Presence of bilateral visual acuity loss from any source
* Inability to demonstrate fixation stability on eye movement monitored testing
* Inability to follow training instructions

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bascom Palmer Eye Institute, University of Miami Health Services, Miami, Florida
  - Flaum Eye Institute, University of Rochester Medical Center, Rochester, New York
  - Scheie Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No subjects were excluded from the study between recruitment and randomization to assigned groups.
Period: Overall Study
Arm/Group | Training in the Blind Field | Training in the Intact Field
Started | 25 | 23
Completed | 23 | 23
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training in the Blind Field | Training in the Intact Field | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.8) | 61.5 (9.4) | 59.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 19 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48
Preliminary deficit size [Mean (Standard Deviation); unit: square degrees of visual angle] — The total area of the subject's deficit, as measured by Humphrey perimetry using a 24-2 testing pattern. This value was calculated by combining testing results from both eyes and interpolating between the tested points to a resolution of 0.1 deg of visual angle. Regions of the visual field with a pattern deviation value (as measured by the Humphrey perimeter) of less than -5 dB were then recorded as part of the deficit. The total area of these combined regions is reported here in square degrees of visual angle.
  square degrees of visual angle | 819.7 (190.6) | 755.2 (167.6) | 788.8 (181.0)
Patients with right sided deficits [Count of Participants; unit: Participants] — Total number of patients with a visual deficit localized to the right hand side of the visual field. The number of patients with a left-side localized deficit is the difference between the total number of subjects and the right-side deficit count.
  Participants | 10 | 10 | 20
Time since lesion [Median (Inter-Quartile Range); unit: months] — The length of time, in months, between the reported date of the stroke that induced visual loss in a patient and their enrollment in the study.
  months | 15.0 [5.7 to 47.3] | 15.5 [6.2 to 57.6] | 15.28 [6.1 to 47.3]

OUTCOME MEASURES:

1. Primary Outcome: 24-2 Humphrey PMD Change From Baseline to 6-month Post-training Timepoint
Description: Change in the perimetric mean deviation (PMD) generated by standard Humphrey automated perimetry using a 24-2 testing pattern between baseline and post-training after a 6-month training interval.
Time Frame: 6 months
Population: All subjects that completed the assigned training were included in analysis. Each eye was analyzed independently for the primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: decibels
Units Other Than Participants: Eyes
Groups:
- Training in the Blind Field (Left Eye); Training in the Blind Field (Right Eye): Training in the blind field using software
  Training in the blind field: A computer software and chin-rest necessary to perform visual training will be loaned to each patient to use at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a pre-determined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. They will train daily (about 40-60 minutes total), 5 to 7 days per week, for at least 24 weeks.
  Final outcomes will be reported independently for Left and Right eyes.
- Training in the Intact Field (Left Eye); Training in the Intact Field (Right Eye): Training in the intact field using software
  Training in the intact field: A computer software and chin-rest necessary to perform visual training will be loaned to each patient to use at home. They will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion of a small cloud of dots located at a pre-determined location in the intact field of vision. The computer program will automatically create a record of patient performance during each home training session. They will train daily (about 40-60 minutes total), 5 to 7 days per week, for at least 24 weeks.
  Final outcomes will be reported independently for Left and Right eyes.
Arm/Group | Training in the Blind Field (Left Eye) | Training in the Intact Field (Left Eye) | Training in the Blind Field (Right Eye) | Training in the Intact Field (Right Eye)
Number analyzed (Participants) | 23 | 23 | 23 | 23
Number analyzed (Eyes) | 23 | 23 | 23 | 23
decibels | 0.84 [0.22 to 1.47] | 0.10 [-0.52 to 0.72] | 0.58 [0.07 to 1.08] | 0.12 [-0.38 to 0.62]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial enrollment and the conclusion of final assessment. For a given subject this period covered approximately 6 months.
Description: Subjects were in open communication with study staff throughout their training period and invited to report any issues if they arose. At the conclusion of training subjects were interviewed and asked to report any adverse events they may have experienced.
Arm/Group | Training in the Blind Field | Training in the Intact Field
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03350919/Prot_SAP_000.pdf